CLINICAL TRIAL: NCT04060758
Title: An Open Label, Comparative, Sequential-dose, Multi-centre Study Involving Intracameral Administration of a PA5108 Latanoprost FA SR Ocular Implant Into the Eye of Patients With Mild-moderate Glaucoma
Brief Title: Open Label, Sequential-dose Study of PA5108 Latanoprost FA SR Ocular Implant for Mild-moderate Glaucoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PolyActiva Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LATA CS102
Record Dates: First submitted 2019-08-05; First posted 2019-08-19 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Open Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 14.7 mcg (single dose) (Experimental): PA5108 Latanoprost FA SR Ocular Implant which releases 14.7 mcg.
  Interventions: Drug: PA5108 Latanoprost FA SR Ocular Implant
- 26.6 mcg (single dose) (Experimental): PA5108 Latanoprost FA SR Ocular Implant which releases 26.6 mcg.
  Interventions: Drug: PA5108 Latanoprost FA SR Ocular Implant
- 35.5 mcg (single dose) (Experimental): PA5108 Latanoprost FA SR Ocular Implant which releases 35.5 mcg.
  Interventions: Drug: PA5108 Latanoprost FA SR Ocular Implant
- 14.7 mcg (repeat dose) (Experimental): Repeat dose of PA5108 Latanoprost FA SR Ocular Implant which releases 14.7 mcg.
  Interventions: Drug: PA5108 Latanoprost FA SR Ocular Implant

INTERVENTIONS:
Drug: PA5108 Latanoprost FA SR Ocular Implant — Ocular Implant
  Other Names: PA5108

SUMMARY:
This is a multi-centre, open label, interventional, comparative, phase I study to identify a safe and efficacious dose (within the range of 14.7mcg to 35.5 mcg) of PA5108 (PolyActiva product code) Latanoprost free acid (FA) sustained release (SR) Ocular Implant in adults who have Primary Open Angle Glaucoma.

DETAILED DESCRIPTION:
This is a multi-centre, open label, interventional, comparative, phase Ib dose ranging study to identify a safe and efficacious dose (within the range of 14.7 to 35.5 microgram) of PA5108 Latanoprost FA SR Ocular Implant in adults who have Primary Open Angle Glaucoma (POAG).

The proposed study is a single ascending dose design to determine the minimum effective dose that provides the target of >20% IOP lowering effect at 12 weeks with minimal adverse events.

Up to three single-dose cohorts will be assessed from the following implant strengths:

* 35.5 microgram
* 26.6 microgram
* 14.7 microgram

In addition, a repeat-dose cohort will be assessed from the following implant strength:

o 14.7 microgram

A first cohort of participants will be recruited and dosed with the 14.7 mcg PA5108 Latanoprost FA SR Ocular Implant. A second cohort of participants will be recruited after SMC review of 6-week data of the first cohort and dosed with the 26.6 mcg PA5108 Latanoprost FA SR Ocular Implant. A third cohort of participants will be recruited after SMC review of 6-week data of the second cohort and repeat-dosed with 14.7 mcg PA5108 Latanoprost FA SR Ocular Implant. A fourth cohort of participants will be recruited and dosed with the 35.5 mcg PA5108 Latanoprost FA SR Ocular Implant

Prior to study registration, participants will have been medicated with intraocular pressure (IOP) lowering drop therapy, including a prostaglandin analogue, to manage their POAG. The IOP lowering drops will be stopped in the intent to treat eye within 29 to 43 days prior to the date of implant administration. Participants will be required to have an unmedicated (post wash-out) 8:00am IOP ≥ 24 mmHg and ≤ 36mmHg in the intent to treat eye at either of two screening visits 2-weeks apart. Additionally, the IOP at 12:00 noon and 4:00 pm must be ≥ 20mmHg and ≤ 36mmHg on the same screening visit where the 8:00am IOP was ≥ 24 mmHg and ≤ 36mmHg.

The PA5108 Latanoprost FA SR Ocular Implant will be administered to one eye (unilateral) of each participant.

IOP will be monitored and if after implant administration is found to rise ≥30% over baseline in the study eye, IOP lowering eye drops will be restarted.

The study will recruit up to 10 participants per cohort/dose level. After screening, eligible participants enrolled in the single-dose cohorts will be administered a single PA5108 Latanoprost FA SR Ocular Implant by clear corneal injection to the anterior chamber of the eye, by means of a custom-built injector fitted with a 27G pre-loaded needle at Day 0. Whereas eligible participants enrolled in the repeat-dose cohort will be administered a single PA5108 Latanoprost FA SR Ocular Implant by clear corneal injection to the anterior chamber of the eye, by means of a custom-built injector fitted with a 27G pre-loaded needle at Day 0, and again at Week 21.

The study will end at the later of Visit 12 (48-weeks) for the last participant in the repeat dose cohort, or when the last of the study implants are no longer visible in the study eye and the IOP in the same eye has returned to a normal clinical care range, or 12-weeks has passed since the implant was no longer visible regardless of IOP.

Participants in the single dose cohorts will attend the study site for follow up on Day 1 post implant administration, and then Week 6, 12, (optionally 15), 18, (optionally 21), 26, 32 and if required subsequent 6-week intervals until the implant has completely biodegraded and the IOP of the same eye has returned to normal clinical care range or 12-weeks has passed since the implant was no longer visible. Implant biodegradation will be confirmed by biomicroscopy and gonioscopy examination at Week 6, 12, optionally 15, 18, optionally 21, 26 & 32, and if necessary, every 6-weeks thereafter.

Participants in the repeat dose cohort will attend the study site for follow up on Day 1 post implant administration, and then Week 6, 12,18, Week 21 (when they will be administered the second dose), Day 1 post repeat dose, Week 27, 33, 42, 48 and if required subsequent 6-week intervals until the implant has completely biodegraded and the IOP of the same eye has returned to normal clinical care range or 12-weeks has passed since the implant was no longer visible. Implant biodegradation will be confirmed by biomicroscopy and gonioscopy examination at Week 6,12,18, 21,27, 33,42 & 48, and if necessary, every 6-weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

Participants who:

* Diagnosis of primary open angle glaucoma.
* Unmedicated 8:00am IOP ≥ 24 mmHg and ≤ 36mmHg in the intent to treat eye. Additionally, the IOP at 12:00 and 16:00 hrs must be ≥ 20mmHg and ≤ 36mmHg.
* Corrected visual acuity in each eye greater than or equal to +0.3logMAR.
* Minimum central endothelial cell density of greater than or equal to 1600 cells per mm2
* Currently managing their POAG with IOP lowering drop therapy.

Exclusion Criteria:

Participants who:

* Have pseudoexfoliation or pigment dispersion component, history of angle closure, or narrow angles.
* Have a history of or current ocular inflammation.
* Have aphakic eyes or only one eye.
* Recent surgery in the study eye surgery (including laser).
* Clinically significant ocular disease in either eye (e.g., corneal oedema, uveitis, severe keratoconjunctivitis sicca or infection) which might interfere with the study.
* Known sensitivity to any component of the product (e.g. latanoprost or polytriazole sensitivity), or to topical therapy used during course of study (e.g. povidone iodine, or anaesthetics).
* Ocular medication in either eye of any kind within 30 days of screening.
* Central corneal thickness in either eye that is less than 470 µm or greater than 630 µm at screening (or a difference between the eyes >70 µm).
* Any abnormality in either eye preventing reliable applanation tonometry, including aphakic eyes or significant corneal guttatae.
* Any other clinically significant disease (as determined by physician) which might interfere with the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2025-05-13 (Actual); Study Completion 2025-05-13 (Actual)

PRIMARY OUTCOMES:
Effective dose | Intraocular Pressure (IOP) change measured at; baseline, week 12 and week 26.
  Determine the minimum effective dose (as daily release rate of LtpFA) that achieves an IOP lowering effect >20% with minimal adverse events.
Safety and Tolerability-incidence of treatment emergent Adverse Events | Incidence of Treatment-Emergent Adverse Events throughout the study (up to 1 year).
  Assess the safety and tolerability of PA5108 Latanoprost FA SR Ocular Implant in adults with Open Angle Glaucoma (Primary). Incidence of Treatment-Emergent Adverse Events from visit 1 until end of study. Safety laboratory evaluations (biochemistry, haematology, urinalysis). Physical examinations and vital signs. Changes in ocular examinations from baseline to end of study.

SECONDARY OUTCOMES:
Ease of Use | At visit 2-Day 0, after use of device to insert the implant into the eye.
  Assess the ease of use of the bespoke administration device- Administering ophthalmologist's assessment of ease of use of the bespoke administration device, verbal communication.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Coote, Principal Investigator — Melbourne Eye Specialists
Locations (9):
- Australia (8):
  - PersonalEYES, Castle Hill, New South Wales
  - Goodwood Eye Centre, Millswood, South Australia
  - Bendigo Eye Clinic, Bendigo, Victoria
  - Centre for Eye Research Australia, East Melbourne, Victoria
  - Essendon Eye Clinic, Essendon, Victoria
  - Melbourne Eye Specialists, Fitzroy, Victoria
  - Eyes First, Springvale, Victoria
  - Eye Surgery Associates, Vermont South, Victoria
- Capital Eye Specialists, Te Aro, New Zealand

IPD SHARING:
Plan to Share IPD: No